CLINICAL TRIAL: NCT03995966
Title: A Clinical Trial for Treatment-Resistant Subtypes of Self-Injurious Behavior
Brief Title: A Clinical Trial for Self-Injurious Behavior
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Louis Hagopian, PhD, Director of the Neurobehavioral Unit, Department of Behavioral Psychology, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00179539
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Self-Injurious Behavior
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: A randomized crossover design will be employed. Specifically, the approach will include using randomly permuted block randomization, stratified by subtype (Subtype 2 or Subtype 3 ASIB). If the treatment based on the first approach is deemed ineffective, a 3-day washout period will occur (where no treatment is applied), followed by the initiation of the second approach to treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subtype 2 Automatically Maintained SIB (Active Comparator)
  Interventions: Behavioral: Noncontingent Reinforcement (NCR); Behavioral: Combination Treatment
- Subtype 3 Automatically Maintained SIB (Active Comparator)
  Interventions: Behavioral: Noncontingent Reinforcement (NCR); Behavioral: Combination Treatment

INTERVENTIONS:
Behavioral: Noncontingent Reinforcement (NCR) — This treatment for ASIB is based on reinforcer competition. Noncontingent Reinforcement (NCR) will consist of first conducting a competing stimulus assessment (CSA) to identify stimuli (toys, massagers, etc.) associated with reductions in ASIB and high levels of engagement. Treatment then involves NCR in which alternative sources of reinforcement are made freely available to compete with reinforcement maintaining ASIB. Providing additional sources of reinforcement is thought to decrease ASIB by producing a shift in the allocation of responding toward accessing the newly available reinforcement. Additional, more restrictive components may be added if the competing stimuli (CS) are ineffective in reducing ASIB. These additional components are applied in accordance to the least-restrictive treatment model and include response blocking, response reduction procedures, protective equipment, or mechanical restraint.
Behavioral: Combination Treatment — Combination Treatment is based on the same principles as NCR, but differs in three ways: 1) It includes three pre-treatment assessments that seek to establish competing stimuli, tasks, and self-control equipment through prompting and reinforcement; ; 2) Intensive training in each of these components is conducted to strengthen skills needed to fully access available reinforcement to compete with ASIB; and 3) Combination treatment is assessed, which includes the noncontingent delivery of competing stimuli and differential reinforcement of alternative behavior to reinforce engagement with competing tasks, and use of alternative self-control equipment. This will increase the amount and vary the sources of alternative reinforcement to more effectively reduce ASIB and self-restraint. Restrictive components may be applied as described for the NCR treatment.

SUMMARY:
At least one quarter of the 18 million persons in the US with intellectual and developmental disabilities engage in self-injurious behavior (SIB), which can result in injuries, disfigurement, and loss of function (e.g., blindness). SIB that persists in the absence of social reinforcement has been referred to as automatically maintained SIB (ASIB). Research has shown that the sensitivity of ASIB to disruption by alternative reinforcement is identifiable in a standardized assessment, predicts response to treatment, and provides a quantifiable basis for subtyping ASIB. This research has also identified two subtypes that are highly resistant to behavioral treatment using reinforcement alone, necessitating the use of protective equipment and other procedures to minimize injury. The proposed study is a clinical trial that will allow systematic comparison of the effectiveness of two behavioral treatments targeting treatment-resistant subtypes of ASIB.

DETAILED DESCRIPTION:
Research shows that automatically maintained self-injurious behavior (ASIB) is comprised of treatment-responsive (Subtype 1) and treatment-resistant subtypes (Subtypes 2 and 3). The primary objective of the clinical trial is to compare two behavioral treatments for the treatment-resistant subtypes of ASIB: Subtypes 2 and 3. Noncontingent Reinforcement (NCR) with competing stimuli (toys that reduce occurrence of SIB) is widely used, but its outcomes are not optimal for most cases with Subtype-2 and -3 ASIB. Noncontingent reinforcement (NCR) includes two phases: 1) Pre-Treatment Assessment to identify competing stimuli and 2) NCR Treatment. Combination Treatment (CT) is based on the same principles as NCR (reinforcer competition), but increases the amount and varies the sources of alternative reinforcement to more effectively reduce ASIB and self-restraint. CT involves the use of competing stimuli, competing tasks (activities that reduce SIB), and self-control training to reduce self-restraint or teach alternative, more adaptive forms of self-control. CT includes three phases: 1) Pre-Treatment Assessments, 2) Intensive Training, and 3) Combination Treatment. Pre-Treatment Assessments will identify competing stimuli, tasks, and self-control equipment; and Intensive Training will strengthen skills needed to fully access available reinforcement to compete with ASIB, and establish self-control skills to replace debilitating self-restraint. Following the Intensive Training phase, CT combines noncontingent access to competing stimuli with differential reinforcement of alternative behavior (DRA) to reinforce engagement with competing tasks, and use of alternative self-control equipment.

Each study participant will be randomly assigned to first receive either NCR or CT using randomly permuted block randomization, stratified by subtype. Each approach includes more than one phase, but both end with a treatment phase. If the first treatment applied is ineffective, based on defined criteria (including the level of improvement and number of treatment sessions), a 3-day washout period will follow where no treatment is applied, and then the second approach will be initiated culminating in the application of that treatment (either NCR or CT).

Following a demonstration of treatment efficacy (for either the first or second treatment that is applied), any additional non-reinforcement treatment components that were added will be withdrawn to determine whether those components remain necessary. If a strong treatment effect does not maintain, the additional components will be reapplied. Treatment generalization will be initiated, and if the effects are maintained the trial will end.

If the first treatment that is applied is effective, that treatment will continue to be applied and generalization will be conducted (and the participant will not crossover to the other treatment approach).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with intellectual disabilities
* Admitted to the Neurobehavioral Unit Inpatient program at the Kennedy Krieger Institute
* Between the ages of 4 to 25 years
* Exhibits either Subtype 2 or 3 automatically maintained self-injurious behavior

Exclusion Criteria:

* Children in foster care
* Non-English speakers
* Individuals with a medical condition that could interfere with participation, or place an individual at increased risk

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-Injurious Behavior (SIB) | Upon recruitment, the study duration for individuals who complete the entire protocol (including receiving both treatments via the crossover design) is anticipated to be between 57 and 92 days.
  Data on self-injurious behavior (SIB) will be collected in real time using direct observation of the behavior. Data will be collected on the frequency of ASIB which will be transformed into responses per minute. Data will be collected during baseline and treatment phases. The primary outcome measure for SIB will include the percentage change in SIB during treatment relative to baseline. Following the completion of the study, statistical analyses will be conducted evaluating the percentage change in SIB and the relative difference in percentage change for each of the treatments.
Self-Restraint | Upon recruitment, the study duration for individuals who complete the entire protocol (including receiving both treatments via the crossover design) is anticipated to be between 57 and 92 days.
  Data on self-restraint will be collected in real time using direct observation of the behavior. Data will be collected on the duration of self-restraint which will be transformed into the percentage of session with self-restraint. Data will be collected during baseline and treatment phases. The primary outcome measure for self-restraint will the absolute duration of self-restraint. Following the completion of the study, statistical analyses will be conducted evaluating the percentage change in the duration self-restraint and the relative difference in percentage change for each of the treatments.

SECONDARY OUTCOMES:
Engagement | Upon recruitment, the study duration for individuals who complete the entire protocol (including receiving both treatments via the crossover design) is anticipated to be between 57 and 92 days.
  Data on engagement with the competing stimuli, competing task, and self-control equipment will be collected in real time using direct observation of the behavior. Data will be collected on the duration of engagement, which will be transformed into the percentage of session with engagement. Data will be collected during control and test stimuli phases of the Pre-Assessments and during baseline and treatment phases of the Treatment. The secondary outcome measure for engagement will include the percentage change during treatment relative to baseline.
Other Problem Behavior (for some participants) | Upon recruitment, the study duration for individuals who complete the entire protocol (including receiving both treatments via the crossover design) is anticipated to be between 57 and 92 days.
  Data on other topographies of problem behavior (e.g., aggression, disruptions) will be collected in real time using direct observation of the behavior. Data will be collected on the frequency of other problem behavior which will be transformed into responses per minute. Data will be collected during baseline and treatment phases. The secondary outcome measure for other problem behavior will include the percentage change during treatment relative to baseline.
Self-Injury Trauma Scale (SITS) | At enrollment; repeated at completion of treatment, anticipated to be between 57 and 92 days from enrollment.
  The Self-Injury Trauma Scale (SITS) measures surface tissue damage. In Section 1: Measurement of Surface Trauma, the number of injuries at each body location is scored (0=no wounds, 1=1 wound, 2=2-4, and 3=5 or more), type of injury (AL = abrasion/laceration, and CT = contusion), and severity of injury (1 = red, irritated, local swelling or discoloration; 2 = superficial break in skin or extensive swelling; 3 = extensive break in skin, avulsion present, chronic wound, disfigurement or tissue rupture). For Section 2: Topography, each type of self-injury the participant exhibits is recorded. For Section 3: Scoring Summary, a Number Index is obtained for the number of injuries across all body locations (0=no injuries, 1=1-4, 2=5-8, 3=9-12, 4=13-16, and 5=17 or more); a Severity Index provides a composite of severity scores (0= no injuries; 1=all 1s; 2=one 2, no 3s, 3 = two or more 2s; 4 = one 3; 5 = two or more 3s); Estimate of Current Risk is recorded as Low, Moderate, or High.

CONTACTS AND LOCATIONS:
Overall Officials: Louis P Hagopian, PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Podlewski J, Opolski M. [Skin carcinoma in a contused head injury treated surgically]. Wiad Lek. 1974 Mar 15;27(6):557-9. No abstract available. Polish. PMID 4830359
- [Background] Canal P, Erill S. Effects of calcium dobesilate upon thurfyl nicotinate erythema in man. J Med. 1971;2(6):375-9. No abstract available. PMID 5292128
- [Background] Hagopian LP, Frank-Crawford MA. Classification of self-injurious behaviour across the continuum of relative environmental-biological influence. J Intellect Disabil Res. 2018 Dec;62(12):1108-1113. doi: 10.1111/jir.12430. Epub 2017 Oct 13. PMID 29027294